STATISTICAL PLAN
Evaluating Alternative Medical Therapies in Primary Hyperparathyroidism
NCT02525796
7/31/2015

## Statistical Plan

<u>Analytic Plan, Sample Size and Power:</u> A sample size of 20 subjects per intervention arm (n=60 total) has been chosen using <u>conservative</u> calculations. The **primary outcome**, ΔPTH in response to randomized drug therapy, will be analyzed using a 2-arm ANOVA analysis evaluating the difference between EPL and placebo. A 3-arm ANOVA including the amiloride arm will also be conducted. Sample size calculations are presented in **Figure** using preliminary data from the RAAS-PARC study where the  $\Delta$ PTH= -13 pg/mL was seen with RAAS inhibition in participants with P-HPTH, but also using a more conservative estimate (-9.0 pg/mL) that is 25% lower. It is expected that  $\Delta$ PTH with placebo will range from 0 to +4.57pg/mL, and calculations have been made to anticipate that amiloride may serve as either a negative control (like placebo) or positive control (like EPL). With these conservative estimates, a sample size of 20 subjects/arm will be sufficient to demonstrate a  $\Delta$ PTH with a type I error of <0.05 and power=80%.

The **secondary outcomes**, change in calcium, will be analyzed in the same fashion as PTH. For calcium, sample size calculations are based on decreases in *total calcium* seen in the RAAS-PARC study ( $\Delta$ Ca= -0.32 mg/dL); treatment with EPL is expected to result in a <u>much greater</u> effect estimate. Thus, using *conservative* estimates of  $\Delta$ Ca= -0.20 to -0.32 mg/dL, a sample size of 20 subjects per intervention arm will be sufficient to achieve 80% power.

**<u>Figure:</u>** Sample size calculations based on  $\Delta PTH$ .

| | ΔΡΤΗ | ΔΡΤΗ | ΔΡΤΗ | SD | Sample Size per Arm | |
|---|---|---|---|---|---|---|
| | Placebo | Amiloride | SPIRO | | PWR=0.8 | PWR=0.9 |
| 2-arms | 0 pg/mL | - | -9.0 pg/mL | 9.4 | 19 | 24 |
| 2-a | 0 pg/mL | - | -13.0 pg/mL | 9.4 | 10 | 13 |
| | 0 pg/mL | 0 pg/mL | -9.0 pg/mL | 9.4 | 17 | 22 |
| S | 0 pg/mL | 0 pg/mL | -13.0 pg/mL | 9.4 | 9 | 11 |
| 3-arms | 0 pg/mL | -6.5 pg/mL | -13.0 pg/mL | 9.4 | 12 | 15 |
| က် | 0 pg/mL | -9.0 pg/mL | -13.0 pg/mL | 9.4 | 11 | 14 |
| | 0 pg/mL | -13.0 pg/mL | -13.0 pg/mL | 9.4 | 9 | 11 |

Figure: Sample size calculation based on  $\Delta Ca$ .

| ΔCa | ΔCa | ΔCa SPIRO | | Sample Si | ze per Arm |
|---------|-----------|-------------|------|-----------|------------|
| Placebo | Amiloride | ACA SPIRO | SD | PWR=0.8 | PWR=0.9 |
| 0 mg/dL | 0 mg/dL | -0.20 mg/dL | 0.21 | 17 | 22 |
| 0 mg/dL | 0 mg/dL | -0.32 mg/dL | 0.21 | 8 | 10 |